CLINICAL TRIAL: NCT02576834
Title: Suicide Prevention Among Substance Abusing Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natasha Slesnick, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014B0532; R34DA037845 (NIH)
Record Dates: First submitted 2015-10-10; First posted 2015-10-15 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTSP + SAU (Experimental): 10 sessions of Cognitive Therapy for Suicide Prevention (CTSP) provided over 6 months, with optional 9 booster sessions + SAU
  Interventions: Behavioral: Cognitive Therapy for Suicide Prevention; Other: Services as Usual
- Services as Usual (SAU) (Other): client receives services they would normally receive within the community
  Interventions: Other: Services as Usual

INTERVENTIONS:
Behavioral: Cognitive Therapy for Suicide Prevention — 10 sessions of cognitive therapy for suicide prevention provided, along with optional 9 booster sessions + SAU
  Other Names: CTSP
  Arms: CTSP + SAU
Other: Services as Usual — Services as usually provided in the community
  Other Names: SAU

SUMMARY:
The literature is characterized by a dearth of information on interventions for homeless youth, and no suicide prevention intervention has been tested with these youth. Such focus is critical as suicide is the leading cause of death among homeless youth. Therefore, this study seeks to address this gap in the research literature with the goal to identify an effective strategy to intervene in suicide ideation in this population.

DETAILED DESCRIPTION:
While research on homeless youth is increasing, there is a dearth of information regarding effective interventions for these youth. This is of significant concern because studies indicate that 70-95% report problem alcohol or drug use and 66% to 89% of homeless youth have a mental health disorder. Suicide is the leading cause of death with up to 68% of youth reporting a lifetime suicide attempt. Among those who have attempted, an average of 6.2 attempts is reported. In addition, lifetime suicide ideation rates have ranged from 14% to 66.5%. Some predictors of suicide among homeless youth have been identified. These include substance use, childhood physical and sexual abuse, victimization experiences while living on the streets, and psychological functioning, including depression, hopelessness, distress tolerance, impulse control, social support, and problem solving. This study uses general cognitive theory, complemented with concepts from two suicide specific theoretical models, to guide our intervention and conceptual change model. Consonant with the pilot R34 announcement, this study's goal is to pilot test an intervention that has previously demonstrated feasibility and promise with adolescent suicide attempters and efficacy with a low-income sample of adults, "The Cognitive Therapy Intervention for Suicide Attempters." One-hundred fifty homeless youth with recent severe suicide ideation will be randomly assigned to the experimental cognitive therapy for suicide prevention (CTSP) + services as usual (SAU) (n=75) or to SAU alone (n=75). SAU includes those services normally offered through a local drop-in center. Follow-up assessments will be conducted at 3, 6, and 9-months post-baseline. It is hypothesized that youth receiving CTSP+SAU will show greater reductions in suicide ideation (primary outcome), substance use and depressive symptoms (secondary outcomes) over time compared to SAU alone. Furthermore, theoretically-derived mediators will be tested to shed light on mechanisms associated with change. The data from this study will be used to determine the initial efficacy of this promising intervention, and determine whether findings warrant a broader scale effectiveness trial. Ultimately, attention towards reducing suicide risk among these youth has the potential to reduce premature mortality, hospitalization and loss of human capital in a very high risk population of youth.

ELIGIBILITY:
Inclusion Criteria:

* 18-24
* meet McKinney Vento definition for homelessness.
* Youth reports at least one episode of severe suicide ideation in the past 90 days.

Exclusion Criteria:

* Evidence of unremitted psychosis or other condition which would impair youth's ability to understand and participate in the research.
* Youth requires psychiatric hospitalization.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
change in suicide ideation | 9 months
  suicide ideation assessed at baseline, 3, 6 and 9 months post-baseline using self-report measures

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Department of Human Development and Family Science, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No